CLINICAL TRIAL: NCT01602588
Title: A Randomised Phase 2 Trial Investigating the Additional Benefit of Hydroxychloroquine(HCQ)to Short Course Radiotherapy (SCRT) in Patients Aged 70 Years and Older With High Grade Gliomas (HGG)
Brief Title: A Randomised Trial Investigating the Additional Benefit of Hydroxychloroquine(HCQ)to Short Course Radiotherapy (SCRT) in Patients Aged 70 Years and Older With High Grade Gliomas (HGG)
Acronym: HCQ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL11/0404
Record Dates: First submitted 2012-05-08; First posted 2012-05-21 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Hydroxychloroquine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Experimental): Patients randomised to Arm B will receive Short Course Radiotherapy plus Hydroxychloroquine 200mg bd from 14 days post surgery until clinical or radiological progression.
  Interventions: Drug: Hydroxychloroquine
- Arm A: SCRT alone (Active Comparator): Patients randomised to Arm A will receive standard treatment of Short Course Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Hydroxychloroquine — 200mg bd from 14 days post surgery until clinical or radiological progression
  Other Names: HCQ
  Arms: Arm B
Radiation: Radiotherapy — Short Course radiotherapy
  Arms: Arm A: SCRT alone

SUMMARY:
There is emerging evidence that hydroxychloroquine (HCQ), a drug used commonly in the prevention/ treatment of malaria, rheumatoid arthritis and lupus erythematosus, may improve survival outcome in a variety of cancers including HGG, with few side effects.

In this trial the investigators wish to investigate whether treatment with radiotherapy and hydroxychloroquine is more effective than treatment with radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥70 yrs identified through the neurooncology MDT.
* A histological diagnosis of HGG, either from biopsy or resection.
* A life expectancy of > 2 months
* An ECOG performance status of 0/1
* Absolute neutrophil count ≥ 1.5 x 109
* Platelet count ≥ 100 x 109
* Bilirubin ≤ 1.5 mg/dL (or ≤ 25.6 µmol/L)
* Creatinine ≤ 2 times upper limit of normal (ULN)
* ALT and AST ≤ 4 times ULN
* Mini Mental Status Exam score ≥ 17 (Appendix 10)
* Written informed consent
* Ready to start radiotherapy within 4 weeks of surgery

Exclusion Criteria:

* Concurrent psoriasis unless the disease is well controlled and patient is under the care of a specialist for the disorder who agrees to monitor for exacerbations
* Prior macular degeneration or diabetic retinopathy
* Concurrent serious infection or medical illness that would preclude study therapy
* Another malignancy within the past 5 years except for curatively treated carcinoma in situ or basal cell carcinoma of the skin
* Porphyria
* Glucose- 6 phosphate dehydrogenase (G6PD) deficiency
* Alcoholic liver disease
* Any other concurrent severe/uncontrolled medical conditions
* Currently taking amiodarone
* Prior radiotherapy, chemotherapy, immunotherapy, biologic agents (e.g., immunotoxins, immunoconjugates, antisense agents, peptide receptor antagonists, interferons, interleukins, tumour-infiltrating lymphocytes, lymphokine-activated killer cell therapy, or gene therapy), or hormonal therapy for brain tumour
* Prior polifeprosan 20 with carmustine implant (Gliadel wafer) or GliaSite® brachytherapy
* Concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
* Other concurrent chemotherapeutic or investigational agents for this cancer (Concurrent glucocorticoids will be allowed
* Documented side effects to chloroquine or related agents.
* Unable to give informed consent
* Patients with a history of a psychological illness or condition that in the opinion of the investigator may adversely affect compliance with study medication

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
1 year Survival | The survival rate will be calculated by the number of patients alive 1 year after entering the trial.
  The primary endpoint of the trial is survival at one year

SECONDARY OUTCOMES:
Toxicity | Toxicity will be assessed during and up to 30 days after treatment
  Adverse Events will be collected for all patients in the trial during treatment and up to 30 days afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Short, Professor, Principal Investigator — St James's University Hospital
Locations (15):
- United Kingdom (15):
  - St James's University Hospital, Leeds, West Yorkshire
  - Glan Clwyd Hospital, Bodelwyddan
  - Addenbrooke's Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - University College Hospital, London
  - Guy's and St Thomas's Hospitals, London
  - Charing Cross Hospital, London
  - Christie Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - Norfolk & Norwich University Hospitals, Norwich
  - The Royal Preston Hospital, Preston
  - Royal Stoke University Hospital, Stoke-on-Trent